CLINICAL TRIAL: NCT05635461
Title: A Randomized, Open-Label, Single Oral Dose, Three-Way Cross-Over Trial to Evaluate the Relative Bioavailability of CVN424 Suspension &Tablet Formulations Including an Assessment of the Effect of Food on the Tablet Formulation in Healthy Adult Volunteers
Brief Title: Relative Bioavailability and Food Effect Study of CVN424
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevance Beta, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cerevance (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CVN424-102
Record Dates: First submitted 2022-11-07; First posted 2022-12-02 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Suspension (fasted) (Active Comparator): 150 milligrams (mg) of CVN424 administered in a single dose of suspension formulation.
  Interventions: Drug: CVN424
- Tablet (fed) (Active Comparator): 150 milligrams (mg) tablet of CVN424 administered in a single dose after ingestion of a standardized high-fat, high-calorie meal according to FDA Guidance for Industry (Food-effect bioavailability and fed bioequivalence studies, Jun 2022).
  Interventions: Drug: CVN424
- Tablet (fasted) (Active Comparator): 150 milligrams (mg) tablet of CVN424 administered in a single dose.
  Interventions: Drug: CVN424

INTERVENTIONS:
Drug: CVN424 — 150 mg of either tablet or suspension formulation

SUMMARY:
This is a Randomized, Open-Label, Single Oral Dose, Three-Way Cross-Over Trial to Evaluate the Relative Bioavailability of CVN424 Suspension and Tablet Formulations in Healthy Volunteers Under Fasted and Fed Conditions.

DETAILED DESCRIPTION:
32 healthy male or female participants will be enrolled in 1 of 6 sequences (designated as 1 through 6, respectively) in an ascending fashion. Sequences 1, 3, 4, and 5 will have 5 participants each, and Sequences 2 and 6 will have 6 participants each.

Each sequence will proceed through the three cross-overs (suspension-fasted, tablet-fed, and tablet-fasted) according to the schematic, with dosing to occur on Days 1 of Periods 1, 2, and 3. Participants in the fasted portion of each sequence will be dosed under overnight fasted conditions and will remain fasted for 4 hours post-dose. Water consumption is permitted as desired except for 1 hour before and after administration of the Study Drug.

To assess the effect of food on CVN424 bioavailability in tablet formulation, the single dose will be administered after ingestion of a standardized high-fat, high-calorie meal according to FDA Guidance for Industry (Food-effect bioavailability and fed bioequivalence studies, Jun 2022).

Participants for all sequences will be admitted to the study unit 1 day prior to dosing and remain in the unit for safety and pharmacokinetics (PK) assessments through 96 hours post-dose. The total confinement period will be 5 nights for each period unless extended at the discretion of the Investigator, e.g., for monitoring and/or management of adverse events (AEs).

Once 96-hour post-dose PK has been collected, participants will be discharged from the unit for the remainder of the washout period and return the day prior for their next scheduled dosing period

ELIGIBILITY:
Inclusion Criteria:

* In the Investigator's opinion, the participant can understand and sign the Informed Consent Form (ICF) and comply with all protocol requirements.
* The participant is male or female adult who is 18 to 55 years of age, inclusive at the time of Screening.
* Participant weighs at least 45 kilograms (kg) (99 pounds [lbs]) and has a BMI between 18.0 and 35.0 kg/m2, inclusive at Screening.
* The participant is medically healthy with no clinically significant (CS) or relevant abnormalities in medical history, physical exam, vital signs, ECG, and laboratory evaluations (hematology, chemistry, and urinalysis) as assessed by the Investigator.
* Female participants of childbearing potential and male participants with female partners of childbearing potential must agree to either remain abstinent or use two methods of adequate and reliable contraception (see Section 9.1.12) throughout the study and at least 12 weeks after the last dose of study drug has been taken.

Exclusion Criteria:

* Vegetarian, Vegan, Lactose intolerant, or follows a Kosher diet.
* Evidence of clinically significant neurologic or other disorder or impairment that, in the opinion of the Investigator, is reasonably expected to impact the ability of the participant to participate or confound the study results.
* A current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, any surgical intervention known to impact absorption [e.g., bariatric surgery or bowel resection]). Note, history of cholecystectomy is permitted if there is no evidence of malabsorption per the Investigator.
* A history of cancer or other malignancy, with the exception of low-grade cervical intraepithelial neoplasia, low-grade (low-risk) prostate cancer, or 5-year cancer-free survivors of basal or squamous cell carcinoma or higher-grade cervical intraepithelial neoplasia or prostate cancer.
* A positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or a human immunodeficiency virus (HIV) infection at Screening.
* Any clinically significant abnormalities in labs: biochemistry (including liver function test [LFT], estimated glomerular filtration rate [eGFR], and glucose), hematology with white blood cell (WBC) differential, c-reactive protein (CRP), coagulation tests, lipase, amylase, albumin, and calcium.
* A supine blood pressure outside the ranges of 80 to 160 mm Hg for systolic and 50 to 100 mm Hg for diastolic, confirmed with up to two repeat tests at the Screening Visit; or symptomatic orthostatic hypotension, in the opinion of the Investigator.
* A resting heart rate outside the range of 40 to 100 beats per minute (bpm) confirmed with up to two repeat tests at the Screening Visit. Note that 40-50 and 90-100 bpm may be permitted only at the discretion of the Investigator.
* Positive urine result for illegal drugs at Screening and Check-In, or history of illicit drug use or alcohol abuse within 1 year prior to the Screening Visit.
* Received any investigational compound (defined as a drug that has not been FDA-approved) within 30 days prior to the first dose of study medication or within 5 half-lives of the investigational compound, whichever is greater.
* Within 14 or 28 days prior to randomization, ingested any of the following excluded medication, supplements, or food products: St. John's wort, ginseng, kava, Ginkgo biloba, Chinese herbs, and melatonin, or known strong inhibitors/inducers of cytochrome P-4503A4/5, including rifampin, clarithromycin, ketoconazole, itraconazole. For full list of prohibited medications and dietary products, (See Table 2 in full protocol).
* Regularly uses nicotine-containing products (including but not limited to cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum). The casual users (≤ 10 cigarettes/week) may participate; however, they must agree to refrain from 30 days before Day 0 (Inpatient Check-in) for the duration of the study or a positive urine cotinine test at Inpatient Check-in.
* Known history of coronary artery disease and hospitalization for myocardial infraction, ischemic heart disease, or congestive heart failure within the 2 years prior to the screening visit.
* Any clinically significant medical, psychiatric, or laboratory abnormality that, in the judgment of the Investigator, is likely to interfere with study participation.
* A history of major depression or risk of suicide according to the Investigator's clinical judgment or has made a suicide attempt.
* Is a study site employee or an immediate family member of a study site employee.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Martin Bexon, MD, Study Chair — Cerevance Beta, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an Open-label, single oral dose, 3-way cross-over trial that evaluated the relative bioavailability of CVN424 suspension and tablet formulations and also included the assessment of the effect of food on the tablet formulation in healthy adult volunteers.
Pre-assignment Details: A total of 32 participants entered the study and were randomized per protocol to 6 treatment sequences.
Groups:
- Treatment Sequence ABC: Participants were randomized to receive single oral dose of CVN424 150 milligrams (mg) on Day 1 of each treatment period in the following sequence: Treatment A: CVN424 150 mg suspension (fasted) in period 1; Treatment B: CVN424 150 mg Tablet (fasted) in period 2 and Treatment C: CVN424 150 mg Tablet (fed) in Treatment period 3. There was a washout period of 14 days between each treatment period.
- Treatment Sequence ACB: Participants were randomized to receive single oral dose of CVN424 150 mg on Day 1 of each treatment period in the following sequence: Treatment A: CVN424 150 mg suspension (fasted) in period 1; Treatment C: CVN424 150 mg Tablet (fed) in Treatment period 2 and Treatment B: CVN424 150 mg Tablet (fasted) in period 3. There was a washout period of 14 days between each treatment period.
- Treatment Sequence BAC: Participants were randomized to receive single oral dose of CVN424 150 mg on Day 1 of each treatment period in the following sequence: Treatment B: CVN424 150 mg Tablet (fasted) in period 1; Treatment A: CVN424 150 mg suspension (fasted) in Treatment period 2 and Treatment C: CVN424 150 mg Tablet (fed) in period 3. There was a washout period of 14 days between each treatment period.
- Treatment Sequence BCA: Participants were randomized to receive single oral dose of CVN424 150 milligrams (mg) on Day 1 of each treatment period in the following sequence: Treatment B: CVN424 150 mg Tablet (fasted) in period 1; Treatment C: CVN424 150 mg Tablet (fed) in period 2 and Treatment A: CVN424 150 mg suspension (fasted) in Treatment period 3. There was a washout period of 14 days between each treatment period.
- Treatment Sequence CAB: Participants were randomized to receive single oral dose of CVN424 150 mg on Day 1 of each treatment period in the following sequence: Treatment C: CVN424 150 mg Tablet (fed) in Treatment period 1; Treatment A: CVN424 150 mg suspension (fasted) in period 2 and Treatment B: CVN424 150 mg Tablet (fasted) in period 3. There was a washout period of 14 days between each treatment period.
- Treatment Sequence CBA: Participants were randomized to receive single oral dose of CVN424 150 mg on Day 1 of each treatment period in the following sequence: Treatment C: CVN424 150 mg Tablet (fed) in Treatment period 1; Treatment B: CVN424 150 mg Tablet (fasted) in period 2 and Treatment A: CVN424 150 mg suspension (fasted) in period 3. There was a washout period of 14 days between each treatment period.
Period: Period 1: Dosing 1 (Day 1)
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 6 | 5 | 6
Completed | 5 | 5 | 5 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 6 | 5 | 6
Completed | 5 | 5 | 5 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Dosing 2 (Day 1)
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 6 | 5 | 6
Completed | 5 | 5 | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period (7 Days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 6 | 4 | 6
Completed | 5 | 5 | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3: Dosing 3 (Day 1)
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 6 | 4 | 6
Completed | 5 | 4 | 5 | 5 | 4 | 6
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Failed Check-In Laboratory | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of all participants who were enrolled and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA | Total
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (9.07) | 36.0 (8.94) | 39.6 (10.11) | 38.2 (7.11) | 37.6 (12.54) | 48.0 (3.29) | 39.6 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 3 | 3 | 3 | 18
  Male | 3 | 1 | 2 | 3 | 2 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 5 | 4 | 2 | 4 | 22
  Not Hispanic or Latino | 2 | 1 | 0 | 2 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 0 | 1 | 0 | 5
  White | 2 | 3 | 5 | 6 | 3 | 5 | 24
  More than one race | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Measured Non Zero Concentration (AUC0-t) of CVN424 Suspension Fasted and Tablet Fasted
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of CVN424 tablet. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set consists of all participants who received study drug and had at least 1 measurable plasma concentration. Only those participants with data available at specified timepoints have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Groups:
- Treatment A: CVN424 150 mg Suspension (Fasted): Participants were randomized to receive single oral dose of 150 mg CVN424 suspension under fasted condition.
- Treatment B: CVN424 150 mg Tablet (Fasted): Participants were randomized to receive a single oral dose of 150 mg CVN424 tablet under fasted condition.
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted)
Number analyzed (Participants) | 30 | 26
Hours*nanograms per milliliter | 16790 (19.3) | 10100 (31.8)
Statistical Analysis 1: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment B: CVN424 150 mg Tablet (Fasted); Test type: Other; Geometric Mean Ratio = 60.13, 90% CI 2-sided [56.12 to 64.42] — Geometric mean ratio was obtained by multiplying 100 with ratio of test (CVN424 tablet fasted) and reference (CVN424 suspension fasted)

2. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 96 Hours (AUC 0-96h) of CVN424 Suspension Fasted and Tablet Fasted
Description: Blood samples were collected at indicated time points for PK analysis of CVN424 tablet. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted)
Number analyzed (Participants) | 30 | 26
Hours*nanograms per milliliter | 16780 (19.3) | 10100 (31.8)
Statistical Analysis 1: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment B: CVN424 150 mg Tablet (Fasted); Test type: Other; Geometric Mean Ratio = 60.12, 90% CI 2-sided [56.12 to 64.42] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of CVN424 Suspension Fasted and Tablet Fasted
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted)
Number analyzed (Participants) | 30 | 26
nanograms per milliliter | 812.9 (28.9) | 231.1 (40.6)
Statistical Analysis 1: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment B: CVN424 150 mg Tablet (Fasted); Test type: Other; Geometric Mean Ratio = 27.94, 90% CI 2-sided [25.09 to 31.13] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Time to Reach Cmax (Tmax) of CVN424 Suspension and Tablet
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Median (Full Range); unit: hours
Groups:
- Treatment C: CVN424 150 mg Tablet (Fed): Participants were randomized to receive a single oral dose of 150 mg CVN424 tablet under fed condition.
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 30 | 26 | 31
hours | 2.040 [1.00 to 3.08] | 3.526 [1.50 to 48.09] | 4.055 [2.05 to 6.07]
Statistical Analysis 1: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment B: CVN424 150 mg Tablet (Fasted); Test type: Other; p < 0.0001, ANOVA; Median Difference (Final Values) = 1.04, 90% CI 2-sided [0.9265 to 2.2470]
Statistical Analysis 2: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; p < 0.0001, ANOVA; Median Difference (Final Values) = 2.78, 90% CI 2-sided [2.4475 to 3.0035]

5. Primary Outcome: Time Taken for Drug to Appear in Systemic Circulation Following Administration (Tlag) of CVN424 Suspension and Tablet
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 30 | 26 | 31
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.51]
Statistical Analysis 1: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment B: CVN424 150 mg Tablet (Fasted); Test type: Other; Median Difference (Final Values) = 0.00, 90% CI 2-sided [0.000 to 0.000]
Statistical Analysis 2: Comparison: Treatment A: CVN424 150 mg Suspension (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; p = 0.0010, ANOVA; Median Difference (Final Values) = 0.25, 90% CI 2-sided [0.0000 to 0.2510]

6. Secondary Outcome: AUC(0-t) of CVN424 Tablet Fed and Tablet Fasted
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 26 | 31
Hours*nanograms per milliliter | 10100 (31.8) | 16340 (20.0)
Statistical Analysis 1: Comparison: Treatment B: CVN424 150 mg Tablet (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; Geometric Mean Ratio = 161.57, 90% CI 2-sided [150.96 to 172.92] — Geometric mean ratio was obtained by multiplying 100 with ratio of test (CVN424 tablet Fed) and reference (CVN424 tablet fasted)

7. Secondary Outcome: AUC(0-96 Hrs) of CVN424 Tablet Fed and Tablet Fasted
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 26 | 31
Hours*nanograms per milliliter | 10100 (31.8) | 16340 (20.0)
Statistical Analysis 1: Comparison: Treatment B: CVN424 150 mg Tablet (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; Geometric Mean Ratio = 161.59, 90% CI 2-sided [150.98 to 172.95] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Cmax of CVN424 Tablet Fed and Tablet Fasted
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 26 | 31
Nanograms per milliliter | 231.1 (40.6) | 693.8 (23.5)
Statistical Analysis 1: Comparison: Treatment B: CVN424 150 mg Tablet (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; Geometric Mean Ratio = 304.19, 90% CI 2-sided [273.51 to 338.31] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Tmax of CVN424 Tablet Fed and Tablet Fasted
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 26 | 31
hours | 3.526 [1.50 to 48.09] | 4.055 [2.05 to 6.07]
Statistical Analysis 1: Comparison: Treatment B: CVN424 150 mg Tablet (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; p = 0.0662, ANOVA; Median Difference (Final Values) = 0.99, 90% CI 2-sided [0.0060 to 1.5370]

10. Secondary Outcome: Tlag of CVN424 Tablet Fed and Tablet Fasted
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60,72, 84 and 96 hours post-dose
Population: PK Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 26 | 31
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.51]
Statistical Analysis 1: Comparison: Treatment B: CVN424 150 mg Tablet (Fasted) vs Treatment C: CVN424 150 mg Tablet (Fed); Test type: Other; p = 0.0039, ANOVA; Median Difference (Final Values) = 0.25, 90% CI 2-sided [0.0000 to 0.2510]

11. Secondary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence in a clinical research study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug.
Time Frame: Up to Day 35
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
Number analyzed (Participants) | 30 | 30 | 32
Participants | 8 | 11 | 11

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: Adverse events were collected in Safety analysis set that consist of all participants who were enrolled and received the study drug.
Arm/Group | Treatment A: CVN424 150 mg Suspension (Fasted) | Treatment B: CVN424 150 mg Tablet (Fasted) | Treatment C: CVN424 150 mg Tablet (Fed)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 8/30 | 11/30 | 11/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: CVN424 150 mg Suspension (Fasted) (N=30) | Treatment B: CVN424 150 mg Tablet (Fasted) (N=30) | Treatment C: CVN424 150 mg Tablet (Fed) (N=32)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 5
Tremor (Nervous system disorders) | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05635461/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05635461/SAP_001.pdf